CLINICAL TRIAL: NCT01143038
Title: A Phase 2 Interventional Single Arm Study Describing Platelet Responses and ITP Remission Rates in Adult Subjects With Immune Thrombocytopenia Purpura Receiving Romiplostim
Brief Title: Interventional Study in Adults With Immune Thrombocytopenia Purpura (ITP) Receiving Romiplostim
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20080435; 2010-019987-35 (EudraCT Number)
Record Dates: First submitted 2010-06-10; First posted 2010-06-14 (Estimated); Results first posted 2016-02-24 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romiplostim (Experimental): Participants received romiplostim administered weekly by subcutaneous injection during the 12-month treatment period. The starting dose was 1 μg/kg with weekly dose increases continued in increments of 1 μg/kg/week to a maximum dose of 10 μg/kg in an attempt to reach a target platelet count of ≥ 50 x 10^9/L.
  Interventions: Biological: Romiplostim

INTERVENTIONS:
Biological: Romiplostim — Romiplostim will be administered weekly by subcutaneous injection
  Other Names: AMG 531; Nplate

SUMMARY:
The purpose of this study is to describe the number of months with a platelet response over a 12 month treatment period and to describe ITP remission rates in adults with ITP receiving romiplostim.

DETAILED DESCRIPTION:
The study includes a 4-week screening period, a 12-month romiplostim treatment period, and a romiplostim dose-tapering period.

During the 12-month treatment period romiplostim doses could be increased or decreased to maintain a platelet count between ≥ 50 x 10^9/L and ≤ 200 x 10^9/L. Participants who dose reduce such that they no longer require treatment with romiplostim during the 12-month treatment period will continue with all required study procedures up to 12 months and will be monitored for ITP remission for at least 6 months.

At the completion of the 12-month treatment period, participants receiving only romiplostim and with a platelet count ≥ 50 x 10^9/L will enter the tapering period, during which the romiplostim dose will be decreased by 1 µg/kg every 2 weeks, for up to 19 weeks. If a participant maintains a platelet count of ≥ 50 x 10^9/L in the absence of romiplostim and all medications for ITP (concomitant or rescue), the participant will be followed for at least 6 months to confirm the incidence of ITP remission. If a participant's platelet count falls below 50 x 10^9/L and the participant has tapered off treatment with romiplostim, the participant will enter the stabilization period and reinitiate romiplostim for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Subject has been diagnosed with primary ITP according to the American Society of Hematology (ASH) guidelines (George et al, 1996) and previously received only 1st line therapies.

First line therapy is defined as corticosteroids, immunoglobulin G (IVIG), anti-D and vinca alkaloids (used for the treatment of ITP related thrombocytopenia only). A platelet transfusion at any time during the six month period since the original diagnosis would not exclude the subject from study participation

* Initial diagnosis of primary ITP within 6 months of enrollment
* Age ≥ 18 years at screening
* A single platelet count ≤ 30 x 10⁹/L at any time during the screening period
* Subject or subject's legally acceptable representative has provided informed consent

Exclusion Criteria:

* Known history of a bone marrow stem cell disorder
* Surgical resection of the spleen
* Subject has a history of cancer or current malignancy other than basal cell carcinoma or cervical cancer in-situ with active treatment or disease within 5 years of screening
* Known history of congenital thrombocytopenia
* Known history of hepatitis B, hepatitis C, or human immunodeficiency virus
* Positive H. pylori by urea breath test or stool antigen test at screening
* Known history of systemic lupus erythematosus, Evans syndrome, or autoimmune neutropenia
* Known history of antiphospholipid antibody syndrome or positive for lupus anticoagulant
* Known history of disseminated intravascular coagulation, hemolytic uremic syndrome, or thrombotic thrombocytopenic purpura
* Previous history of recurrent venous thromboembolism or thrombotic events or an occurrence within 5 years of enrollment.
* Previous use of romiplostim, pegylated recombinant human megakaryocyte growth and development factor (PEG-rHuMGDF), eltrombopag, recombinant human thrombopoietin (rHuTPO) or any platelet producing agent
* Rituximab (for any indication) or mercaptopurine (6-MP) or anticipated use during the time of the proposed study
* All hematopoietic growth factors including interleukin-11 (IL-11) (oprelvekin) within 4 weeks before the screening visit
* Alkylating agents use at any time before or during the screening visit or anticipated during the time of the proposed study
* Known hypersensitivity to any recombinant E. coli-derived product (eg, Infergen, Neupogen, Somatropin, and Actimmune)
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational agent(s)
* Subject will have any other investigational procedures performed while enrolled in this clinical study
* Subject is pregnant or breast feeding, or planning to become pregnant within 5 weeks after the end of treatment
* Female subject of child bearing potential is not willing to use, in combination with her partner, highly effective contraception during treatment and for 4 weeks after the end of treatment
* Subject has previously enrolled into a romiplostim study
* Subject will not be available for protocol required study visits, to the best of the subject's and investigator's knowledge
* Subject has any kind of disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2013-09-20 (Actual); Study Completion 2013-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (45):
- United States (8):
  - Research Site, Anaheim, California
  - Research Site, Orange, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Bethesda, Maryland
  - Research Site, Hickory, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Richlands, Virginia
- Australia (3):
  - Research Site, Randwick, New South Wales
  - Research Site, Woolloongabba, Queensland
  - Research Site, Adelaide, South Australia
- Czechia (3):
  - Research Site, Brno
  - Research Site, Ostrava-Poruba
  - Research Site, Prague
- France (5):
  - Research Site, Bondy
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Pessac
  - Research Site, Toulouse
- Germany (4):
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Düsseldorf
- Italy (8):
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Monza (MB)
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Roma
  - Research Site, San Giovanni Rotondo FG
  - Research Site, Vicenza
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Wroclaw
- Spain (5):
  - Research Site, Málaga, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Alcorcón, Madrid
  - Research Site, Majadahonda, Madrid
- United Kingdom (4):
  - Research Site, Coventry
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Oxford

REFERENCES:
- [Background] Newland A, Godeau B, Priego V, Viallard JF, Lopez Fernandez MF, Orejudos A, Eisen M. Remission and platelet responses with romiplostim in primary immune thrombocytopenia: final results from a phase 2 study. Br J Haematol. 2016 Jan;172(2):262-73. doi: 10.1111/bjh.13827. Epub 2015 Nov 5. PMID 26537623
- [Background] Cines DB, Wasser J, Rodeghiero F, Chong BH, Steurer M, Provan D, Lyons R, Garcia-Chavez J, Carpenter N, Wang X, Eisen M. Safety and efficacy of romiplostim in splenectomized and nonsplenectomized patients with primary immune thrombocytopenia. Haematologica. 2017 Aug;102(8):1342-1351. doi: 10.3324/haematol.2016.161968. Epub 2017 Apr 14. PMID 28411254
- [Background] Kuter DJ, Newland A, Chong BH, Rodeghiero F, Romero MT, Pabinger I, Chen Y, Wang K, Mehta B, Eisen M. Romiplostim in adult patients with newly diagnosed or persistent immune thrombocytopenia (ITP) for up to 1 year and in those with chronic ITP for more than 1 year: a subgroup analysis of integrated data from completed romiplostim studies. Br J Haematol. 2019 May;185(3):503-513. doi: 10.1111/bjh.15803. Epub 2019 Feb 21. PMID 30793285
- [Background] Kuter DJ, Arnold DM, Rodeghiero F, Janssens A, Selleslag D, Bird R, Newland A, Mayer J, Wang K, Olie R. Safety and efficacy of self-administered romiplostim in patients with immune thrombocytopenia: Results of an integrated database of five clinical trials. Am J Hematol. 2020 Jun;95(6):643-651. doi: 10.1002/ajh.25776. Epub 2020 Mar 21. PMID 32129511
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ninety-eight adults with immune thrombocytopenia purpura (ITP) were screened for the study; 23 were considered screen failures. Seventy-five participants were enrolled at 32 study centers in Australia, the European Union, and North America from 30 November 2010 to 21 September 2012.
Pre-assignment Details: The study included a 12-month romiplostim treatment period, and a romiplostim dose-tapering period. Participants who maintained a platelet count of ≥ 50 x 10^9/L in the absence of romiplostim and all medications for ITP (concomitant or rescue) were followed for at least 6 months to confirm the incidence of ITP remission.
Groups:
- Romiplostim: Participants received romiplostim administered weekly by subcutaneous injection during the 12-month treatment period. The starting dose was 1 μg/kg with weekly dose increases in increments of 1 μg/kg/week to a maximum dose of 10 μg/kg to reach a target platelet count of ≥ 50 x 10^9/L. At the completion of the 12-month treatment period, participants receiving only romiplostim and with a platelet count ≥ 50 x 10^9/L entered the tapering period, during which the romiplostim dose was decreased by 1 µg/kg every 2 weeks, for up to 19 weeks. Participants who had tapered off treatment with romiplostim and whose platelet count dropped below 50 x 10^9/L could reinitiate romiplostim for up to 8 weeks.
Period: Overall Study
Arm/Group | Romiplostim
Started | 75
Completed | 59 (Defined as completion of romiplostim treatment)
Not Completed | 16
Not completed — Withdrawal by Subject | 4
Not completed — Requirement for alternative therapy | 5
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 2
Not completed — Protocol Deviation | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Romiplostim
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 31
Race [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Black (or African American) | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 72
  Other | 0
  Unknown | 1
Ethnicity [Number; unit: participants]
  Hispanic/Latino | 6
  Not Hispanic/Latino | 69
Time since ITP diagnosis [Median (Full Range); unit: months] | 2.2 [0.1 to 6.6]
Platelet Count at Screening [Mean (Standard Deviation); unit: x 10^9/L] | 19.78 (15.80)

OUTCOME MEASURES:

1. Primary Outcome: Number of Months With Platelet Response During the 12-Month Treatment Period
Description: The primary endpoint was the number of months a participant achieved a platelet response during the 12-month treatment period. A platelet response for any 1 month was defined as the median of platelet counts measured in the month ≥ 50 x 10^9/L. Platelet counts within 4 weeks following a rescue medication use or following splenectomy were considered non-response. Months without any platelet count measurement were considered as months with no platelet response.
Time Frame: 12 months
Population: Safety Analysis Set includes all participants who received at least 1 dose of romiplostim.
Measure: Mean (Standard Error); unit: months
Arm/Group | Romiplostim
Number analyzed (Participants) | 75
months | 9.2 (0.4)
Statistical Analysis 1: Comparison: Romiplostim; Test type: Superiority or Other; Mean = 9.2, 95% CI 2-sided [8.3 to 10.1] — Based on the t-distribution
Statistical Analysis 2: Comparison: Romiplostim; Bootstrap analysis; Test type: Superiority or Other; Bootstrap mean = 9.1, 95% CI 2-sided [8.3 to 10.0], Standard Error of Mean 0.4 — Estimates are based on bootstrap method with 1000 samples with replacement

2. Secondary Outcome: Percentage of Participants With ITP Remission
Description: ITP remission was defined as maintaining every platelet count ≥ 50 x 10^9/L for at least 6 months in the absence of romiplostim and any other therapies to treat ITP.
Time Frame: Up to 24 months
Population: Safety analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 75
percentage of participants | 32.0 [21.7 to 43.8]

3. Secondary Outcome: Percentage of Participants With Splenectomy During the 12-month Treatment Period
Description: If treatment with romiplostim was deemed ineffective or intolerable by the investigator, a splenectomy may have been performed.
Time Frame: 12 months
Population: Safety analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 75
percentage of participants | 1.3 [0.0 to 7.2]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. The event does not necessarily have a causal relationship with study treatment. A serious adverse event is defined as an adverse event that meets at least one of the following serious criteria: • fatal • life threatening • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • congenital anomaly/birth defect • other significant medical hazard. Whether an adverse event was treatment-related (TRAE) or not was determined by investigator.
Time Frame: From first dose date of romiplostim to end of study (up to 24 months).
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 75
participants
  All adverse events | 63
  Serious adverse events | 17
  Leading to discontinuation of romiplostim | 4
  Leading to discontinuation from study | 3
  Fatal adverse events | 0
  Treatment-related adverse event | 21
  Treatment-related serious adverse events | 3
  TRAE leading to discontinuation of romiplostim | 2
  TRAE leading to discontinuation from study | 2
  Treatment-related fatal adverse events | 0

5. Secondary Outcome: Number of Participants Who Developed Antibodies to Romiplostim
Description: The number of participants who developed antibody formation (defined as negative at baseline and positive at post-baseline, transient or persistent) to romiplostim, endogenous thrombopoietin (eTPO), and thrombopoietin mimetic peptide (TMP, the peptide component of romiplostim) was summarized.
Time Frame: Baseline and at end of treatment (based on response to treatment, this could occur between 12 months and approximately 18 months)
Population: Safety analysis set participants with available results
Measure: Number; unit: participants
Arm/Group | Romiplostim
Number analyzed (Participants) | 69
participants
  Antibodies to romiplostim | 2
  Antibodies to TPO | 1
  Antibodies to TMP | 2
  Neutralizing antibodies to romiplostim | 1
  Neutralizing antibodies to TPO | 0
  Neutralizing antibodies to TMP | 0

ADVERSE EVENTS:
Time Frame: From first dose date of romiplostim to end of study (up to 24 months).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Romiplostim
Serious Adverse Events (participants affected / at risk) | 17/75
Other Adverse Events (participants affected / at risk) | 50/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=75)
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Erysipelas (Infections and infestations) | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 1
Transaminases Increased (Investigations) | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Reversible Ischaemic Neurological Deficit (Nervous system disorders) | 1
Delirium Tremens (Psychiatric disorders) | 1
Renal Failure Acute (Renal and urinary disorders) | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Dapsone Syndrome (Skin and subcutaneous tissue disorders) | 1
Peripheral Vascular Disorder (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=75)
Vertigo (Ear and labyrinth disorders) | 4
Conjunctivitis (Eye disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 5
Fatigue (General disorders) | 6
Influenza (Infections and infestations) | 7
Nasopharyngitis (Infections and infestations) | 10
Rhinitis (Infections and infestations) | 4
Upper Respiratory Tract Infection (Infections and infestations) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Petechiae (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Haematoma (Vascular disorders) | 8
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.